CLINICAL TRIAL: NCT00493961
Title: The Effects of 7 Days of Exogenous Pulsatile GnRH Treatment on the Pituitary-Gonadal Axis in Hypogonadotropic Hypogonadal Subjects
Brief Title: Studying the Effects of 7 Days of Gonadotropin Releasing Hormone (GnRH) Treatment in Men With Hypogonadism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, Harvard Reproductive Endocrine Sciences Center, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: U54HD028138-447; U54HD028138 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Kallmann Syndrome; Idiopathic Hypogonadotropic Hypogonadism; GnRH Deficiency
Keywords: Kallmann Syndrome; Idiopathic Hypogonadotropic Hypogonadism; GnRH deficiency
MeSH Terms: conditions — Kallmann Syndrome; Idiopathic Hypogonadotropic Hypogonadism | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gonadotropin releasing hormone (GnRH) — Pulsatile GnRH (25 ng/kg per bolus every two hours via microinfusion pump)

SUMMARY:
Men with Idiopathic Hypogonadotropic Hypogonadism (IHH) lack a hormone called gonadotropin releasing hormone (GnRH). This hormone is important for starting puberty, maintaining testosterone levels, and fertility. The purpose of this study is to research the effects of treating IHH men with GnRH for 7 days.

DETAILED DESCRIPTION:
Despite variability in the triggers, timing, and pace of sexual maturity between species, all species utilize the final pathway of hypothalamic secretion of gonadotropin releasing hormone (GnRH) to initiate and maintain the reproductive axis. Thus, GnRH is required for reproductive competence in the human. The classic studies from the 1970s clearly demonstrate that pulsatile release of GnRH from the hypothalamus is a prerequisite for physiologic gonadotrope function. Absence, decreased frequency or decreased amplitude of pulsatile GnRH release results in the clinical syndrome of hypogonadotropic hypogonadism (HH). The phenotypic expression of GnRH deficiency in the human demonstrates considerable heterogeneity. Defining the physiology of GnRH is critical to understanding the clinical heterogeneity of isolated GnRH deficiency and its comparison to other conditions resulting in hypogonadotropic hypogonadism (HH). The overall goal of this protocol is to investigate the neuroendocrine control of reproduction and specifically the physiology and pathophysiology of GnRH secretion and action in the human male.

Subjects will be selected from a group of adult men (18-65 years)based on the demonstration of a low testosterone level (<100 ng/dL) in association with low or inappropriately normal gonadotropin levels. All patients will undergo an initial assessment that includes an overnight 12-hour frequent blood sampling study to determine their degree of endogenous GnRH secretion. Following the overnight evaluation, subjects will have daily outpatient visits for 7 consecutive days when they will receive a GnRH bolus followed by 2hrs of blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic hypogonadotropic hypogonadism (IHH) or Kallmann syndrome (KS)Adult male 18-65 years of age
* Serum testosterone <100 ng/dL

Exclusion Criteria:

* No specific exclusion criteria

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1999-01; Primary Completion 2009-11-17 (Actual); Study Completion 2009-11-17 (Actual)

PRIMARY OUTCOMES:
testosterone | daily for 7 days
LH | frequent sampling for 2 hours
FSH | frequent sampling for 2 hours
Inhibin B | daily for 7 days
free alpha subunit | daily for 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Seminara B Stephanie, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Belchetz PE, Plant TM, Nakai Y, Keogh EJ, Knobil E. Hypophysial responses to continuous and intermittent delivery of hypopthalamic gonadotropin-releasing hormone. Science. 1978 Nov 10;202(4368):631-3. doi: 10.1126/science.100883.
- [Background] Seminara SB, Hayes FJ, Crowley WF Jr. Gonadotropin-releasing hormone deficiency in the human (idiopathic hypogonadotropic hypogonadism and Kallmann's syndrome): pathophysiological and genetic considerations. Endocr Rev. 1998 Oct;19(5):521-39. doi: 10.1210/edrv.19.5.0344. No abstract available. PMID 9793755
- [Background] Arimura A, Kastin AJ, Gonzalez-Barcena D, Siller J, Weaver RE, Schally AV. Disappearance of LH-releasing hormone in man as determined by radioimmunoassay. Clin Endocrinol (Oxf). 1974 Oct;3(4):421-5. doi: 10.1111/j.1365-2265.1974.tb02812.x. No abstract available. PMID 4609640
- [Background] Pimstone B, Epstein S, Hamilton SM, LeRoith D, Hendricks S. Metabolic clearance and plasma half disappearance time of exogenous gonadotropin releasing hormone in normal subjects and in patients with liver disease and chronic renal failure. J Clin Endocrinol Metab. 1977 Feb;44(2):356-60. doi: 10.1210/jcem-44-2-356. PMID 320223
- [Background] Clarke IJ, Cummins JT. The temporal relationship between gonadotropin releasing hormone (GnRH) and luteinizing hormone (LH) secretion in ovariectomized ewes. Endocrinology. 1982 Nov;111(5):1737-9. doi: 10.1210/endo-111-5-1737. No abstract available. PMID 6751801
- [Background] Karsch FJ, Bowen JM, Caraty A, Evans NP, Moenter SM. Gonadotropin-releasing hormone requirements for ovulation. Biol Reprod. 1997 Feb;56(2):303-9. doi: 10.1095/biolreprod56.2.303. PMID 9116125
- [Background] Spratt DI, O'Dea LS, Schoenfeld D, Butler J, Rao PN, Crowley WF Jr. Neuroendocrine-gonadal axis in men: frequent sampling of LH, FSH, and testosterone. Am J Physiol. 1988 May;254(5 Pt 1):E658-66. doi: 10.1152/ajpendo.1988.254.5.E658. PMID 3129947
- [Background] Hayes FJ, McNicholl DJ, Schoenfeld D, Marsh EE, Hall JE. Free alpha-subunit is superior to luteinizing hormone as a marker of gonadotropin-releasing hormone despite desensitization at fast pulse frequencies. J Clin Endocrinol Metab. 1999 Mar;84(3):1028-36. doi: 10.1210/jcem.84.3.5579. PMID 10084591
- [Background] Hoffman AR, Crowley WF Jr. Induction of puberty in men by long-term pulsatile administration of low-dose gonadotropin-releasing hormone. N Engl J Med. 1982 Nov 11;307(20):1237-41. doi: 10.1056/NEJM198211113072003. PMID 6813732
- [Background] Whitcomb RW, Crowley WF Jr. Clinical review 4: Diagnosis and treatment of isolated gonadotropin-releasing hormone deficiency in men. J Clin Endocrinol Metab. 1990 Jan;70(1):3-7. doi: 10.1210/jcem-70-1-3. No abstract available. PMID 2403572
- [Background] Filippi G. Klinefelter's syndrome in Sardinia. Clinical report of 265 hypogonadic males detected at the time of military check-up. Clin Genet. 1986 Oct;30(4):276-84. PMID 3791676
- [Background] Fromantin M, Gineste J, Didier A, Rouvier J. [Impuberism and hypogonadism at induction into military service. Statistical study]. Probl Actuels Endocrinol Nutr. 1973 May 3;16:179-99. No abstract available. French. PMID 4147392
- [Background] Filicori M, Butler JP, Crowley WF Jr. Neuroendocrine regulation of the corpus luteum in the human. Evidence for pulsatile progesterone secretion. J Clin Invest. 1984 Jun;73(6):1638-47. doi: 10.1172/JCI111370. PMID 6427277
- [Background] Narasimha Rao P, Moore PH Jr. Synthesis of new steroid haptens for radioimmunoassay. Part I. 15beta-Carboxyethylmercaptotestosterone-bovine serum albumin conjugate. Measurement of testosterone in male plasma without chromatography. Steroids. 1976 Jul;28(1):101-9. doi: 10.1016/0039-128x(76)90129-x. PMID 960143
- [Background] Groome NP, Illingworth PJ, O'Brien M, Pai R, Rodger FE, Mather JP, McNeilly AS. Measurement of dimeric inhibin B throughout the human menstrual cycle. J Clin Endocrinol Metab. 1996 Apr;81(4):1401-5. doi: 10.1210/jcem.81.4.8636341.
- [Background] Landy H, Schneyer AL, Whitcomb RW, Crowley WF Jr. Validation of highly specific and sensitive radioimmunoassays for lutropin, follitropin, and free alpha subunit in unextracted urine. Clin Chem. 1990 Feb;36(2):340-4. PMID 2105862
- [Result] Pitteloud N, Thambundit A, Dwyer AA, Falardeau JL, Plummer L, Caronia LM, Hayes FJ, Lee H, Boepple PA, Crowley WF Jr. Role of seminiferous tubular development in determining the FSH versus LH responsiveness to GnRH in early sexual maturation. Neuroendocrinology. 2009;90(3):260-8. doi: 10.1159/000245383. Epub 2009 Oct 15. PMID 19829004
- [Result] Sykiotis GP, Hoang XH, Avbelj M, Hayes FJ, Thambundit A, Dwyer A, Au M, Plummer L, Crowley WF Jr, Pitteloud N. Congenital idiopathic hypogonadotropic hypogonadism: evidence of defects in the hypothalamus, pituitary, and testes. J Clin Endocrinol Metab. 2010 Jun;95(6):3019-27. doi: 10.1210/jc.2009-2582. Epub 2010 Apr 9. PMID 20382682
- See also: Clinical research studies of the Reproductive Endocrine Unit at the Massachusetts General Hospital. Click here for more information about this study: Effects of Seven Days of Exogenous Pulsatile GnRH Treatment... — http://www.massgeneral.org/reproendo/pages/reu_study_subject.htm